CLINICAL TRIAL: NCT03323996
Title: Impact of a Training in Therapeutic Education on the Relation Between Care Givers and Their Patients
Acronym: METIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2016/307
Record Dates: First submitted 2017-10-25; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Cancer of Liver; Diabetes
MeSH Terms: conditions — Liver Neoplasms; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health Professionals: Health Professionals attending a training in therapeutic education
  Interventions: Other: Semi-Structured interviews
- Patients: Patients of the health Professionals recruited for the study
  Interventions: Other: Semi-Structured interviews

INTERVENTIONS:
Other: Semi-Structured interviews — individual semi-structured interviews

SUMMARY:
This study aims to describe the impact of a training in therapeutic education on the relation between a caregiver and his/her patients.

Subjects are recruited among health professionals attending a training in therapeutic education. Then they are asked to identify up to 5 of their patients to be contacted by the researcher for an interview.

Individual semi-structured interviews are conducted with 20 duo "caregivers / patients" before the training, 1 month and 6 months after the training.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate to 3 interviews

Exclusion Criteria:

* Not fluent French speaker
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health professionnals attending a training in therapeuthic education and their patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Semi-Structured interviews | 9 months
  Qualitative analysis - theorical saturation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No